CLINICAL TRIAL: NCT01911780
Title: An Eight-week Randomised Double-blind Study to Compare the Efficacy and Safety of Telmisartan 80 mg and Amlodipine 5 mg and Hydrochlorothiazide 12.5 mg vs. Telmisartan 80 mg and Hydrochlorothiazide 12.5 mg in Patients With Hypertension Who Fail to Respond Adequately to Treatment With Telmisartan 80 mg and Hydrochlorothiazide 12.5 mg, Followed by a 52 Weeks Extension Study to Assess Long Term Safety of Telmisartan 80 mg and Amlodipine 5 mg and Hydrochlorothiazide 12.5 mg
Brief Title: Compare Efficacy and Safety of Telmisartan/Hydrochlorothiazide With Telmisartan/Hydrochlorothiazide Plus Amlodipine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1348.2
Record Dates: First submitted 2013-07-26; First posted 2013-07-30 (Estimated); Results first posted 2016-03-28 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Hydrochlorothiazide; Amlodipine

ARMS (2):
- telmisartan + HCTZ + amlodipine (Experimental): telmisartan 80 mg + hydrochlorothiazide (HCTZ) 12.5 mg fixed dose combination (FDC) and amlodipine 5 mg capsule (after the 8-week double-blind period, patients will continue the 52-week open label extension period taking 1 telmisartan 80 mg and hydrochlorothiazide 12.5 FDC tablet and 1 amlodipine 5 mg tablet)
  Interventions: Drug: telmisartan + HCTZ; Drug: amlodipine
- telmisartan + HCTZ + placebo (Active Comparator): telmisartan 80 mg + HCTZ FDC tablet and placebo matching amlodipine 5 mg capsule (after the 8-week double-blind period, patients will continue the 52-week open label extension period taking 1 telmisartan 80 mg and hydrochlorothiazide 12.5 FDC tablet and 1 amlodipine 5 mg tablet)
  Interventions: Drug: placebo; Drug: telmisartan + HCTZ

INTERVENTIONS:
Drug: placebo — placebo matching amlodipine capsule
  Arms: telmisartan + HCTZ + placebo
Drug: telmisartan + HCTZ — FDC tablet
  Arms: telmisartan + HCTZ + placebo
Drug: telmisartan + HCTZ — FDC tablet
  Arms: telmisartan + HCTZ + amlodipine
Drug: amlodipine — capsule
  Arms: telmisartan + HCTZ + amlodipine

SUMMARY:
This is a multi-centre, randomised, double-blind, active-controlled, parallel-group comparative trial to compare the fixed dose combination (FDC) of telmisartan 80 mg + hydrochlorothiazide 12.5 mg and amlodipine 5 mg (T80/A5/H12.5 mg) to telmisartan 80 mg+ hydrochlorothiazide 12.5 mg (T80/H12.5 mg) in blood pressure lowering effect at week 8, the end of the double-blind period in essential hypertensive patients who fail to respond adequately to telmisartan 80 mg+ hydrochlorothiazide 12.5 mg.

Patients are assigned to one of the two groups after a 6-week open-label run-in period taking T80/H12.5 mg.

In addition the long-term safety of telmisartan 80 mg+ amlodipine 5 mg+ hydrochlorothiazide 12.5 mg will be evaluated in a 52-week extension period.

In the 52-week open label extension period patients who are assigned to the T80/A5/H12.5 mg group continue the T80/A5/H12.5 mg therapy, and patients who are assigned to the T80/ /H12.5 mg group change to the T80/A5/H12.5 mg therapy.

ELIGIBILITY:
Inclusion criteria:

1. Essential hypertensive patients who have already taking 2 or 3 antihypertensive drugs and mean seated diastolic blood pressure (DBP) must be >=90 and <=114 mmHg and mean seated systolic blood pressure (SBP) must be =<200 mmHg
2. Able to stop all current antihypertensive drugs (other than study medication) from Visit 1b through the end of the trial without risk to the patient based on the investigator's opinion
3. Age 20 years or older

Exclusion criteria:

1. Patients with known or suspected secondary hypertension
2. Patients with clinically relevant cardiac arrhythmia
3. Congestive heart failure with New York Heart Association (NYHA) functional class III-IV
4. Patients with recent cardiovascular events
5. Patients with recent stroke events
6. Patients with a history of sudden deterioration of renal function with angiotensin II receptor blockers or angiotensin converting enzyme inhibitors; or patients with post-renal transplant or post-nephrectomy
7. Patients with hepatic and/or renal dysfunction
8. Pre-menopausal women who are nursing or pregnant

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2013-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (17):
- Japan (17):
  - 1348.2.020 Boehringer Ingelheim Investigational Site, Chiyoda-ku, Tokyo
  - 1348.2.008 Boehringer Ingelheim Investigational Site, Chuo-ku, Fukuoka, Fukuoka
  - 1348.2.018 Boehringer Ingelheim Investigational Site, Chuo-ku,Kobe, Hyogo
  - 1348.2.006 Boehringer Ingelheim Investigational Site, Chuo-ku,Tokyo
  - 1348.2.013 Boehringer Ingelheim Investigational Site, Chuo-ku,Tokyo
  - 1348.2.021 Boehringer Ingelheim Investigational Site, Chuo-ku,Tokyo
  - 1348.2.012 Boehringer Ingelheim Investigational Site, Hirakata, Osaka
  - 1348.2.011 Boehringer Ingelheim Investigational Site, Kasaoka, Okayama
  - 1348.2.001 Boehringer Ingelheim Investigational Site, Kawasaki, Kanagawa
  - 1348.2.019 Boehringer Ingelheim Investigational Site, Kita-ku, Osaka-shi, Osaka
  - 1348.2.014 Boehringer Ingelheim Investigational Site, Kiyota-ku, Sapporo-shi, Hokkaido
  - 1348.2.002 Boehringer Ingelheim Investigational Site, Kumamoto, Kumamoto
  - 1348.2.007 Boehringer Ingelheim Investigational Site, Nakano-ku,Tokyo
  - 1348.2.009 Boehringer Ingelheim Investigational Site, Nishi-ku, Fukuoka, Fukuoka
  - 1348.2.005 Boehringer Ingelheim Investigational Site, Takatsuki, Osaka
  - 1348.2.016 Boehringer Ingelheim Investigational Site, Uji, Kyoto
  - 1348.2.010 Boehringer Ingelheim Investigational Site, Yoshikawa, Saitama

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 239 enrolled patients, 205 patients were entered in the run-in period and 132 were randomized. The remaining 107 patients were withdrawn from the trial before the randomization.
Pre-assignment Details: An eight-week randomised, double-blind study with active-control and parallel-group comparison in Japanese patients plus 52 week extension period.
Groups:
- Telmisartan + HCTZ + Amlodipine: telmisartan 80 mg + hydrochlorothiazide (HCTZ) 12.5 mg fixed dose combination (FDC) and amlodipine 5 mg capsule orally, once daily (after the 8-week double-blind period, patients will continue the 52-week open label extension period taking 1 telmisartan 80 mg and hydrochlorothiazide 12.5 FDC tablet and 1 amlodipine 5 mg tablet)
- Telmisartan + HCTZ + Placebo: telmisartan 80 mg + HCTZ FDC tablet and placebo matching amlodipine 5 mg capsule orally, once daily (after the 8-week double-blind period, patients will continue the 52-week open label extension period taking 1 telmisartan 80 mg and hydrochlorothiazide 12.5 FDC tablet and 1 amlodipine 5 mg tablet)
Period: Double-blind Period (8 Weeks)
Arm/Group | Telmisartan + HCTZ + Amlodipine | Telmisartan + HCTZ + Placebo
Started | 68 | 64
Completed | 65 | 61
Not Completed | 3 | 3
Not completed — Adverse Event | 1 | 2
Not completed — Consent withdrawn not due to AEs | 1 | 1
Not completed — Personal reason | 1 | 0
Period: Extension Period (52 Weeks)
Arm/Group | Telmisartan + HCTZ + Amlodipine | Telmisartan + HCTZ + Placebo
Started | 65 | 61
Completed | 61 | 58
Not Completed | 4 | 3
Not completed — Adverse Event | 3 | 0
Not completed — Consent withdrawn not due to AEs | 0 | 2
Not completed — Personal reason | 1 | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS) was defined as a collection of patients i) randomised to the double-blind period; ii) taking at least 1 dose of either T80/A5/H12.5 mg or T80/H12.5 mg during the double-blind period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Telmisartan + HCTZ + Amlodipine | Telmisartan + HCTZ + Placebo | Total
Number analyzed (Participants) | 68 | 64 | 132
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.1 (10.2) | 54.4 (7.9) | 55.2 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 55 | 49 | 104

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Seated DBP at Trough After 8 Weeks of the Double-blind Period.
Description: Change from baseline in mean seated diastolic blood pressure (DBP) at trough (24-hour post dosing) after 8 weeks of the double-blind period. The results are presented as 'change' rather than 'reduction' i.e., reductions are expressed with negative values'. The 'adjusted mean' is shown as 'mean'.
Time Frame: baseline and 8 weeks
Population: Full analysis set (FAS) was, conforming to the intent-to-treat principle, defined as all patients i) included in the treated set; and ii) taking measurements of seated DBP at reference baseline and at 1 or more time points during the double-blind period
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Telmisartan + HCTZ + Amlodipine | Telmisartan + HCTZ + Placebo
Number analyzed (Participants) | 67 | 64
mmHg | -8.8 (0.8) | -1.3 (0.8)
Statistical Analysis 1: Comparison: Telmisartan + HCTZ + Amlodipine vs Telmisartan + HCTZ + Placebo; Test type: Superiority or Other; p < 0.0001, LOCF-ANCOVA; Last observation carried forward (LOCF) was used as the imputation method; Adjusted mean, comparison = -7.5, 95% CI 2-sided [-9.7 to -5.3], Standard Error of Mean 1.1 — Model includes baseline DBP as a linear covariate, and treatment and center as fixed effects

2. Secondary Outcome: Change From Baseline in Mean Seated SBP at Trough After 8 Weeks of the Double-blind Period.
Description: Change from baseline in mean seated systolic blood pressure (SBP) at trough after 8 weeks of the double-blind period. The results are presented as 'change' rather than 'reduction' i.e., reductions are expressed with negative values'. The 'adjusted mean' is shown as 'mean'.
Time Frame: baseline and 8 weeks
Population: FAS
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Telmisartan + HCTZ + Amlodipine | Telmisartan + HCTZ + Placebo
Number analyzed (Participants) | 67 | 64
mmHg | -10.6 (1.4) | -2.1 (1.5)
Statistical Analysis 1: Comparison: Telmisartan + HCTZ + Amlodipine vs Telmisartan + HCTZ + Placebo; Test type: Superiority or Other; p < 0.0001, LOCF-ANCOVA — Additional information, the p-value is not adjusted for multiplicity; Adjusted mean, comparison = -8.6, 95% CI 2-sided [-12.7 to -4.5], Standard Error of Mean 2.1 — Model includes baseline SBP as a linear covariate, and treatment and center as fixed effects

3. Secondary Outcome: The Percentage of Patients With DBP<90 mmHg and SBP<140 mmHg Blood Pressure at Trough After 8 Weeks of Double-blind Period.
Description: The percentage of patients with DBP<90 mmHg and SBP<140 mmHg as seated blood pressure at trough after 8 weeks of the double-blind period. The results are presented as 'change' rather than 'reduction' i.e., reductions are expressed with negative values'. The 'adjusted mean' is shown as 'mean'.
Time Frame: Double-blind and 8 weeks
Population: FAS
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | Telmisartan + HCTZ + Amlodipine | Telmisartan + HCTZ + Placebo
Number analyzed (Participants) | 67 | 64
Participants | 44.8 [32.6 to 57.4] | 21.9 [12.5 to 34.0]
Statistical Analysis 1: Comparison: Telmisartan + HCTZ + Amlodipine vs Telmisartan + HCTZ + Placebo; Test type: Superiority or Other; p = 0.0052, Regression, Logistic — Additional information, the p-value is not adjusted for multiplicity; Non-completers considered failures (NCF) was used as the imputation method; Odds Ratio (OR) = 3.1, 95% CI 2-sided [1.4 to 7.1] — Exact 95 % confidence interval by Clopper and Pearson. Logistic regression includes treatment and center

4. Secondary Outcome: The Number of Patients With DBP<90 mmHg and SBP<140 mmHg Blood Pressure at Trough After 52 Weeks of Extension Period.
Description: The number of patients with DBP<90 mmHg and SBP<140 mmHg as seated blood pressure at trough after 52 weeks of the extension period. Note, week 52 of the extension period corresponds to 60 weeks after the reference baseline.
  The results are presented as 'change' rather than 'reduction' i.e., reductions are expressed with negative values'. The 'adjusted mean' is shown as 'mean'.
Time Frame: Reference baseline (week 0) and week 60 (end of extension period)
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Telmisartan + HCTZ + Amlodipine | Telmisartan + HCTZ + Placebo
Number analyzed (Participants) | 65 | 61
Participants
  Yes | 41 [32.6 to 57.4] | 33 [12.5 to 34.0]
  No | 24 | 28

5. Secondary Outcome: Change From Baseline in Mean DBP Pressure at Trough After 52 Weeks of the Extension Period.
Description: Change from baseline in mean seated diastolic blood pressure at trough after 52 weeks of the extension period. Note, week 52 of the extension period corresponds to 60 weeks after the reference baseline.
  The results are presented as 'change' rather than 'reduction' i.e., reductions are expressed with negative values'. The 'adjusted mean' is shown as 'mean'.
Time Frame: Reference baseline (week 0) and week 60 (end of extension period)
Population: FAS in the extension period (FASEX OC) was defined as a collection of patients i) included in the FAS; ii) taking at least 1 dose of T80/A5/H12.5 mg in the extension period; and iii) taking measurements of seated DBP at reference baseline and at 1 or more time points in the extension period.
Measure: Mean (Standard Error); unit: mmHg
Groups:
- Telmisartan + HCTZ + Amlodipine + Ext: telmisartan 80 mg + hydrochlorothiazide (HCTZ) 12.5 mg fixed dose combination (FDC) and amlodipine 5 mg capsule orally, once daily (after the 8-week double-blind period, patients will continue the 52-week open label extension period taking 1 telmisartan 80 mg and hydrochlorothiazide 12.5 FDC tablet and 1 amlodipine 5 mg tablet)
- Telmisartan + HCTZ + Placebo + Ext: telmisartan 80 mg + HCTZ FDC tablet and placebo matching amlodipine 5 mg capsule orally, once daily (after the 8-week double-blind period, patients will continue the 52-week open label extension period taking 1 telmisartan 80 mg and hydrochlorothiazide 12.5 FDC tablet and 1 amlodipine 5 mg tablet)
Arm/Group | Telmisartan + HCTZ + Amlodipine + Ext | Telmisartan + HCTZ + Placebo + Ext
Number analyzed (Participants) | 61 | 58
mmHg
  Mean | -11.4 (1.0) | -10.0 (1.0)
  Adjusted mean | -10.9 (1.0) | -10.5 (1.0)
Statistical Analysis 1: Comparison: Telmisartan + HCTZ + Amlodipine + Ext vs Telmisartan + HCTZ + Placebo + Ext; Test type: Superiority or Other; mixed-effects model repeated measures; Adjusted Mean = -0.4, 95% CI 2-sided [-3.1 to 2.3], Standard Error of Mean 1.4 — As a linear covariate, and treatment and visit, treatment by visit interaction and baseline value by visit interaction as fixed effects

6. Secondary Outcome: Change From Baseline in Mean Seated SBP at Trough After 52 Weeks of the Extension Period.
Description: Change from baseline in mean seated systolic blood pressure at trough after 52 weeks of the extension period. Note, week 52 of the extension period corresponds to 60 weeks after the reference baseline.
  The results are presented as 'change' rather than 'reduction' i.e., reductions are expressed with negative values'. The 'adjusted mean' is shown as 'mean'.
Time Frame: Reference baseline (week 0) and week 60 (end of extension period)
Population: FASEX (OC)
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Telmisartan + HCTZ + Amlodipine + Ext | Telmisartan + HCTZ + Placebo + Ext
Number analyzed (Participants) | 61 | 58
mmHg
  Mean | -14.8 (1.6) | -14.3 (1.6)
  Adjusted mean | -13.6 (1.3) | -15.9 (1.4)
Statistical Analysis 1: Comparison: Telmisartan + HCTZ + Amlodipine + Ext vs Telmisartan + HCTZ + Placebo + Ext; Test type: Superiority or Other; mixed-effects model repeated measures; Adjusted Mean = 2.3, 95% CI 2-sided [-1.5 to 6.1], Standard Error of Mean 1.9 — Model includes baseline SBP as a linear covariate, and treatment and visit, treatment by visit interaction and baseline value by visit interaction as fixed effects

ADVERSE EVENTS:
Time Frame: Up to 60 weeks
Groups:
- Telmisartan + HCTZ + Amlodipine - Double Blind Period: Telmisartan 80 mg + hydrochlorothiazide (HCTZ) 12.5 mg fixed dose combination (FDC) and amlodipine 5 mg capsule orally, once daily for 8 weeks (double blind period)
- Telmisartan + HCTZ + Placebo - Double Blind Period: Telmisartan 80 mg + HCTZ FDC tablet and placebo matching amlodipine 5 mg capsule orally, once daily for 8 weeks (double-blind period)
- Telmisartan + HCTZ + Amlodipine - Extension Period: Patients in the 52-week open label extension period taking 1 telmisartan 80 mg and hydrochlorothiazide 12.5 FDC tablet and 1 amlodipine 5 mg tablet who previously received telmisartan 80 mg + hydrochlorothiazide (HCTZ) 12.5 mg fixed dose combination (FDC) and amlodipine 5 mg capsule orally, once daily for 8 weeks in the double blind period. Adverse events which occurred in extension period were collected.
- Telmisartan + HCTZ + Placebo - Extension Period: Patients in the 52-week open label extension period taking 1 telmisartan 80 mg and hydrochlorothiazide 12.5 FDC tablet and 1 amlodipine 5 mg tablet who previously received telmisartan 80 mg + HCTZ FDC tablet and placebo matching amlodipine 5 mg capsule orally, once daily for 8 weeks in the double-blind period. Adverse events which occurred in extension period were collected.
Arm/Group | Telmisartan + HCTZ + Amlodipine - Double Blind Period | Telmisartan + HCTZ + Placebo - Double Blind Period | Telmisartan + HCTZ + Amlodipine - Extension Period | Telmisartan + HCTZ + Placebo - Extension Period
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/64 | 2/65 | 2/61
Other Adverse Events (participants affected / at risk) | 7/68 | 6/64 | 26/65 | 16/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telmisartan + HCTZ + Amlodipine - Double Blind Period (N=68) | Telmisartan + HCTZ + Placebo - Double Blind Period (N=64) | Telmisartan + HCTZ + Amlodipine - Extension Period (N=65) | Telmisartan + HCTZ + Placebo - Extension Period (N=61)
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Lacunar infarction (Nervous system disorders) | 0 | 0 | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Telmisartan + HCTZ + Amlodipine - Double Blind Period (N=68) | Telmisartan + HCTZ + Placebo - Double Blind Period (N=64) | Telmisartan + HCTZ + Amlodipine - Extension Period (N=65) | Telmisartan + HCTZ + Placebo - Extension Period (N=61)
Nasopharyngitis (Infections and infestations) | 6 | 6 | 23 | 16
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.